CLINICAL TRIAL: NCT01460147
Title: Bone and Joint Health in an Adult Hemophilia Population
Brief Title: Osteoporosis and MRI Study in Hemophilia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 001001
Record Dates: First submitted 2011-10-20; First posted 2011-10-26 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Bone Mineral Density; Hemophilia A; Hemophilia B
Keywords: Hemophilia
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Absorptiometry, Photon; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DXA scan + MRI (Other)
  Interventions: Other: DXA scan + MRI

INTERVENTIONS:
Other: DXA scan + MRI — This is a non-drug study. Subjects will receive a dual-energy X-ray absorptiometry (DXA) scan (in the main osteoporosis study) and will undergo magnetic resonance imaging (in the MRI substudy).

SUMMARY:
The purpose of this study is to evaluate bone mineral density in adult subjects with hemophilia versus a comparator population without hemophilia (non-hemophilia age- and gender-matched database) by using the following diagnostic means: dual-energy X-ray absorptiometry (DXA) scanning, clinical scales, quality of life (QOL) scales and biomarkers. In addition to this osteoporosis study, hemophilic arthropathy of the knee with respect to loss of knee cartilage will also be explored by using magnetic resonance imaging (MRI substudy). No investigational product will be dispensed.

ELIGIBILITY:
Inclusion Criteria:

* Male and at least 25 years old at the time of screening
* Moderately severe or severe hemophilia A or B (factor VIII or factor IX <= 2% by chart documentation)
* Ambulatory (ie, not wheel chair dependent)
* Performance status - ECOG of 0 or 1 (= out of bed at least 75% of time)
* Willing and able to comply with the requirements of the protocol and is able to give informed consent

Additional inclusion criteria for MRI Substudy:

* Baseline knee joint space width is >= 3mm at the medial or lateral aspect of either knee as measured by weightbearing fixed flexion PA X-ray
* Able to undergo 1.5 or 3T MRI

Exclusion Criteria:

* Inability to position properly for DXA
* Presence of orthopedic hardware or other artifact in the lumbar spine (L1-L4) or either proximal femur
* Prior documentation of being HIV positive
* Radiosynovectomy or surgical synovectomy within the last 6 months
* Current or past treatment with bone active drugs
* Long-term corticosteroid use [defined as 7.5-mg prednisone daily (or equivalent) for >= 3 months]
* If subject is family member or employee of the investigator

Additional exclusion criteria for MRI Substudy:

* Any contraindication or relative contraindication to MRI
* Less than 3mm knee joint space width at the medial and lateral aspect of both knees on baseline X-ray evaluation
* Knee bleed within 30 days of informed consent
* Prior total knee arthroplasty (TKA)

Min Age: 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-10-30 (Actual); Primary Completion 2012-04-13 (Actual); Study Completion 2012-04-13 (Actual)

PRIMARY OUTCOMES:
Baseline Endpoint: Z-Score by dual-energy X-ray absorptiometry (DXA) at baseline | Baseline
Longitudinal Endpoint: Change in bone mineral density by DXA over 2 years | 2 years
Longitudinal Endpoint: Rate of loss of knee cartilage parameters over 2 years by MRI | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Los Angeles Orthopedic Hospital, Los Angeles, California, United States